CLINICAL TRIAL: NCT05251571
Title: Efficacy of Video-Based Balance and Coordination Exercises in Individuals With Stroke
Brief Title: The Efficiency of Video-Based Exercises in Individuals With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGE2
Record Dates: First submitted 2022-01-31; First posted 2022-02-22 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Stroke
Keywords: Stroke; Telerehabilitation; Balance; Coordination
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Exercise Group with Telerehabilitation (Active Comparator): Exercises such as muscle strengthening exercises applied to antigravity muscles, agonist antagonist spastic muscles, stretching exercises for spastic muscles, weight transfer will be applied, and a telerehabilitation platform will be used in the home exercise program.
  Interventions: Other: Conventional Exercise Group with Telerehabilitation
- Balance Coordination Group with Telerehabilitation (Experimental): Sit and stand exercise from chair, standing posture, weight transfer to right and left extremities, stepping over obstacles, standing on one leg with support from the table, standing on two legs with support from the table, hip abduction with support from the table, extension, flexion, supported tandem walking exercises such as stepping on the stairs, standing functional stretches will be applied. Whatsapp application-based Telerehabilitation platform will be used to deliver the home exercise program.
  Interventions: Other: Balance Coordination Group with Telerehabilitation

INTERVENTIONS:
Other: Conventional Exercise Group with Telerehabilitation — Exercises such as conventional muscle strengthening and stretching given with telerehabilitation are applied.
  Arms: Conventional Exercise Group with Telerehabilitation
Other: Balance Coordination Group with Telerehabilitation — Functional muscle strengthening, stretching, balance and coordination exercises given with telerehabilitation are applied.
  Arms: Balance Coordination Group with Telerehabilitation

SUMMARY:
The aim of the study is to compare the video-based balance coordination exercise program and the video-based conventional exercise program in patients with subacute stroke.

DETAILED DESCRIPTION:
Thanks to telerehabilitation, it will be possible for individuals to learn the exercise programs in the most appropriate way and to communicate easily with their physiotherapists with video images. In this way, it will be ensured that individuals can perform their exercises at the optimum level in non-clinical environments. The aim of the study is to compare the conventional home exercise program performed with video-based telerehabilitation and the balance coordination program in subacute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 40 - 65 years
* Having been diagnosed with stroke by a specialist physician and at least 3 months and maximum 6 months have passed since the diagnosis
* No serious medical complications
* Being able to understand verbal and visual commands
* Getting at least 24 points on the mini mental state test
* Able to walk at least 10 m without assistance using crutches or a walker
* Having signed the consent form

Exclusion Criteria:

* Situations that will prevent assessments or communication with the individual
* Being on psychotropic medication
* People with ataxia or any other cerebellar symptoms
* Other problems that would preclude evaluation and/or treatment

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
FES-I | Change from Baseline FES-I at 6 weeks
  There are 16 items in FES-I that assess the fear of falling during daily activities. FES-I is scored from 0 to 64. Higher scores indicate higher concerns about falling.
ABC | Change from Baseline ABC at 6 weeks
  This scale includes 16 tasks related to indoor and outdoor activities of daily living to measure balance confidence in the elderly with various levels of function. Higher scores indicate more confidence. ABC is scored from 0 to 100. Higher scores indicate higher function.
SSEQ | Change from Baseline SSEQ at 6 weeks
  The 13-item SSEQ is used to measure participants' self-efficacy levels in performing daily functional activities and self-management. SSEQ is scored from 0 to 130. Higher scores indicate higher confidence.

SECONDARY OUTCOMES:
TSQ | Change from Baseline TSQ at 6 weeks
  This questionnaire consists of 14 items. The level of satisfaction of the patients with the software or system from which they receive treatment or other remote rehabilitation services is evaluated. TSQ is scored from 14 to 170. Higher scores indicate higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Özkeskin, PhD, Principal Investigator — Ege University; İsmet Tümtürk, MSc, Principal Investigator — Ege University; Bedriye Karaman, MD, Principal Investigator — Ege University
Locations (1):
- Ege University Hospital Neurology Polyclinic, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No